CLINICAL TRIAL: NCT01871428
Title: A Multicenter, Randomized, Doubleblind, Placebo-Controlled, Phase III Study to Assess the Efficacy, Safety and Tolerability of Aleglitazar Monotherapy Compared With Placebo in Patients With Type 2 Diabetes Mellitus (T2D) Who Are Drug-Naïve to Antihyperglycemic Therapy
Brief Title: A Study of Aleglitazar in Monotherapy in Patients With Type 2 Diabetes Mellitus Who Are Drug-Naïve to Anti-Hyperglycemic Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YC28037
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — aleglitazar

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Aleglitazar (Experimental)
  Interventions: Drug: aleglitazar
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: aleglitazar — 150 mcg orally daily
  Arms: Aleglitazar
Drug: placebo — matching aleglitazar placebo orally daily
  Arms: Placebo

SUMMARY:
This multicenter, randomized, double-blind, placebo-controlled study will evaluate the efficacy, safety and tolerability of aleglitazar monotherapy in patients with Type 2 diabetes mellitus who are drug-naïve to anti-hyperglycemic therapy. Patients will be randomized to receive either aleglitazar 150 mcg orally daily or placebo for 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, >/= 18 years of age
* Diagnosis of Type 2 diabetes mellitus within 12 months prior to screening
* Drug-naïve (defined as no anti-hyperglycemic medication for at least 12 weeks prior to screening and for not longer than 3 consecutive months at any time in the past)
* HbA1c >/= 7% and </= 9.5% at screening or within 4 weeks prior to screening and at pre-randomization visit
* Fasting plasma glucose </= 13.3 mmol/L (</= 240 mg/dL) at pre-randomization visit
* Agreement to maintain diet and exercise habits implemented during the run-in phase during the full course of the study

Exclusion Criteria:

* Pregnant women, women intending to become pregnant during the study period, currently lactating women, or women of child-bearing potential not using highly effective, medically approved birth control methods
* Diagnosis or history of:

  1. Type 1 diabetes mellitus, diabetes resulting from pancreatic injury, or secondary forms of diabetes
  2. Acute metabolic diabetic complications such as ketoacidosis or hyperosmolar coma within the past 6 months
* Any previous treatment with thiazolidinedione or with a dual peroxisome proliferator activated receptor (PPAR) agonist
* Any body weight lowering or lipoprotein-modifying therapy (e.g. fibrates) within 12 weeks prior to screening with the exception of stable (>= 1 month) statin therapy
* Prior intolerance to fibrate
* Triglycerides (fasting) > 4.5 mmol/L (> 400 mg/dL) at screening or within 4 weeks prior to screening
* Clinically apparent liver disease
* Anemia at or within 4 weeks prior to screening
* Inadequate renal function
* Symptomatic congestive heart failure New York Heart Association (NYHA) Class II-IV at screening
* Myocardial infarction, acute coronary syndrome or transient ischemic attack/stroke within 6 months prior to screening visit
* Known macular edema at screening or prior to screening visit
* Diagnosed and/or treated malignancy (except for basal cell skin cancer, in situ carcinoma of the cervix, or in situ prostate cancer) within the past 5 years
* Uncontrolled hypertension
* History of active substance abuse (including alcohol) within the past 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | from baseline to Week 26

SECONDARY OUTCOMES:
Change in lipids | from baseline to Week 26
Change in fasting plasma glucose (FPG) | from baseline to Week 26
Responder rates, defined as target HbA1c: < 7.0%, < 6.5% at Week 26 | 26 weeks
Change in homeostatic index of insulin sensitivity (by Homeostasis Model Assessment for Insulin Sensitivity [HOMA-IS]) | from baseline to Week 26
Change in homeostatic index of beta cell function (by HOMA-BFC) | from baseline to Week 26
Change in markers of insulin sensitivity/cardiovascular risk | from baseline to Week 26
Safety: Incidence of adverse events | approximately 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- China (4):
  - Chongqing
  - Shanghai
  - Shiyan
  - Suzhou
- Hong Kong, Hong Kong
- Malaysia (2):
  - Alor Star
  - Perak